CLINICAL TRIAL: NCT04481984
Title: Effectiveness of a Home-based, Self-administered Exercise Program for Hands in Patients With Systemic Sclerosis: a Randomized Controlled, Single-blind, Clinical Trial
Brief Title: Effectiveness of a Home-based, Self-administered Exercise Program for Hands in Patients With Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Neslihan Gokcen, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cukurova Uni. Neslihan G.
Record Dates: First submitted 2020-07-12; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Systemic Sclerosis; Scleroderma; Hand Rheumatism; Rehabilitation
Keywords: Systemic sclerosis; Scleroderma; Hand; Rehabilitation; Exercise therapy; Self-management
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled, Single-blind, Clinical Study
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The training including isometric and stretching hand exercise was applied once by a physiatrist. A hand exercise ball was used for isometric exercise. Patients performed both stretching exercises and isometric exercises according to the training and printed materials. The home-based exercise program was implemented 7 days per week during an 8-week period. In addition, patients received recommendations such as avoiding cold exposure and trauma.
  Interventions: Other: Home-based Hand exercise
- Control group (Other): Patients received care advice including avoiding cold exposure and trauma.
  Interventions: Other: Care advice

INTERVENTIONS:
Other: Home-based Hand exercise — Isometric exercise; patients squeezed a hand exercise ball for 60 seconds. This exercise repeated 15-times/3 set per day.
  Stretching exercises; self-administered stretching exercises were as follows; i) forearm supination and pronation, ii) wrist flexion and extension, iii) finger flexion, extension, and abduction iv) thumb flexion, extension, and abduction. These exercises repeated 10-times/2 set per day.
  Other Names: Rehabilitation
  Arms: Exercise group
Other: Care advice — Patients received care advice including avoiding cold exposure and trauma.
  Arms: Control group

SUMMARY:
Systemic sclerosis (SSc) is a heterogeneous autoimmune disease characterized by fibrosis of the skin and internal organs. Hand involvement is one of the most observed musculoskeletal involvements in patients with SSc, which can impact on general health, quality of life, and psychological status. Hand exercise programs can help patients to improve not only hand function but also general health status; nevertheless, further randomized control trials (RCTs) are needed to clarify its effect. Hence, the investigators aimed to investigate the effectiveness of home-based, self-administered exercise program for hands in patients with SSc and demonstrate the improvements in general health status.

DETAILED DESCRIPTION:
The current study was designed as a single-blind, prospective, randomized controlled, comparative study with a 2-month follow-up period, conducted in a rheumatology outpatient clinic of a university hospital, between July 2016-June 2019. Female patients with SSc who fulfilled the 2013 ACR/EULAR classification criteria for systemic sclerosis were included in the study. Patients with neurological disorders, arthritis, myositis, amputation of fingers, serious contracture resisting handgrip, and history of undergoing hand surgery were excluded from the study. Patients were enrolled in the study after they signed the written informed consent. Following the assessment of patients in terms of eligibility, patients were randomized into an exercise and a control group. The computerized block randomization method was used to randomize subjects into groups. Both groups were informed about systemic sclerosis and they received the printed materials that include recommendations such as avoiding cold and trauma. The treatment group participated in a single hand exercise training (isometric hand exercise and self-administered stretching) applied by a physiatrist. They additionally received the printable instructions for exercises. Compliance was assessed by a checklist, which included all information on how to exercise and how many times to do them. The investigators aimed to investigate the impact of hand exercise program on hand function and demonstrate its influence on health status, quality of life, and psychological status of patients with SSc.

ELIGIBILITY:
Inclusion Criteria:

- Female systemic sclerosis patients who fulfilled the 2013 ACR/EULAR classification criteria for systemic sclerosis

Exclusion Criteria:

* Patients with neurological disorders,
* Arthritis,
* Myositis,
* Amputation of fingers,
* Serious contracture resisting hand grip
* History of undergoing hand surgery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with Systemic sclerosis
Enrollment: 50 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Handgrip strength | Before treatment to 8 weeks
  Handgrip strength was measured by hydraulic hand dynamometer (JAMAR®,USA) according to the standard protocol, which calculates the average of three consecutive measurements of the dominant hand. The measurements were recorded as kilograms (kg).

SECONDARY OUTCOMES:
Duruoz Hand Index | Before treatment to 8 weeks
  Duruoz Hand Index (DHI) is the 18-item questionnaire assessing hand skill in the kitchen, during dressing, while performing personal hygiene, while performing office tasks, and other general performances. Each item is rated from 0 (no difficulty) to 5 (impossible to do). The sum of the scores varies between 0 and 90. Higher scores indicate the impaired hand function.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Saricam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD may be shared with other researches
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Up to 6 months
Access Criteria: Researchers who would like to access to individual participant data will be reviewed and approved by the principal investigator.

REFERENCES:
- [Background] Landim SF, Bertolo MB, Marcatto de Abreu MF, Del Rio AP, Mazon CC, Marques-Neto JF, Poole JL, de Paiva Magalhaes E. The evaluation of a home-based program for hands in patients with systemic sclerosis. J Hand Ther. 2019 Jul-Sep;32(3):313-321. doi: 10.1016/j.jht.2017.10.013. Epub 2017 Dec 1. PMID 29198478
- [Background] Stefanantoni K, Sciarra I, Iannace N, Vasile M, Caucci M, Sili Scavalli A, Massimiani MP, Passi L, Maset L, Riccieri V. Occupational therapy integrated with a self-administered stretching program on systemic sclerosis patients with hand involvement. Clin Exp Rheumatol. 2016 Sep-Oct;34 Suppl 100(5):157-161. Epub 2016 Apr 14. PMID 27087678
- [Background] Mugii N, Hasegawa M, Matsushita T, Kondo M, Orito H, Yanaba K, Komura K, Hayakawa I, Hamaguchi Y, Ikuta M, Tachino K, Fujimoto M, Takehara K, Sato S. The efficacy of self-administered stretching for finger joint motion in Japanese patients with systemic sclerosis. J Rheumatol. 2006 Aug;33(8):1586-92. PMID 16881115
- [Background] Vannajak K, Boonprakob Y, Eungpinichpong W, Ungpansattawong S, Nanagara R. The short-term effect of gloving in combination with Traditional Thai Massage, heat, and stretching exercise to improve hand mobility in scleroderma patients. J Ayurveda Integr Med. 2014 Jan;5(1):50-5. doi: 10.4103/0975-9476.128859. PMID 24812476
- [Background] Liem SIE, Vliet Vlieland TPM, Schoones JW, de Vries-Bouwstra JK. The effect and safety of exercise therapy in patients with systemic sclerosis: a systematic review. Rheumatol Adv Pract. 2019 Dec 9;3(2):rkz044. doi: 10.1093/rap/rkz044. eCollection 2019. PMID 31858074
- [Background] Rannou F, Boutron I, Mouthon L, Sanchez K, Tiffreau V, Hachulla E, Thoumie P, Cabane J, Chatelus E, Sibilia J, Roren A, Berezne A, Baron G, Porcher R, Guillevin L, Ravaud P, Poiraudeau S. Personalized Physical Therapy Versus Usual Care for Patients With Systemic Sclerosis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2017 Jul;69(7):1050-1059. doi: 10.1002/acr.23098. Epub 2017 Jun 7. PMID 27696703
- [Background] Piga M, Tradori I, Pani D, Barabino G, Dessi A, Raffo L, Mathieu A. Telemedicine applied to kinesiotherapy for hand dysfunction in patients with systemic sclerosis and rheumatoid arthritis: recovery of movement and telemonitoring technology. J Rheumatol. 2014 Jul;41(7):1324-33. doi: 10.3899/jrheum.130912. Epub 2014 Jun 1. PMID 24882841
- [Background] Schouffoer AA, Ninaber MK, Beaart-van de Voorde LJ, van der Giesen FJ, de Jong Z, Stolk J, Voskuyl AE, Scherptong RW, van Laar JM, Schuerwegh AJ, Huizinga TW, Vlieland TP. Randomized comparison of a multidisciplinary team care program with usual care in patients with systemic sclerosis. Arthritis Care Res (Hoboken). 2011 Jun;63(6):909-17. doi: 10.1002/acr.20448. PMID 21312348
- [Derived] Gokcen N, Badak SO, Sarpel T, Sertdemir Y, Erken E. The Efficacy of a Home-Based, Self-Administered Hand Exercise Program for Patients With Systemic Sclerosis: A Randomized Controlled, Evaluator-Blind, Clinical Trial. J Clin Rheumatol. 2022 Mar 1;28(2):e422-e429. doi: 10.1097/RHU.0000000000001752. PMID 34030163

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT04481984/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT04481984/ICF_001.pdf